CLINICAL TRIAL: NCT00628355
Title: Local Injection of Lidocaine Versus Ischemic Compression in Treatment of Woman With Chronic Pelvic Pain Caused by Abdominal Myofascial Pain Syndrome: Randomized Clinical Trial.
Brief Title: Lidocaine Injection and Ischemic Compression on Chronic Pelvic Pain Treatment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lidocaine injection group showed significant improvement in pain
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Omero Benedicto Poli Neto, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCRP10272/2007
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Pelvic Pain
Keywords: lidocaine; ischemic compression; chronic pelvic pain; myofascial pain syndrome
MeSH Terms: conditions — Pelvic Pain; Myofascial Pain Syndromes | interventions — Lidocaine; Acupressure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lidocaine injection (Experimental): Lidocaine injection. Women randomized for this treatment was submitted to 2 milliliters of lidocaine 0,5% without vasoconstrictor, directly and perpendicularly on trigger point.
  Patients received lidocaine injections once a week for 4 weeks
  Interventions: Drug: lidocaine
- Ischemic compression (Experimental): Women randomized for treatment with ischemic compression will be first subjected to transcutaneal electrostimulation (TENS) for 30 minutes on trigger point to inhibit the painful stimulation. For this will be used 100 Hertz of frequency and pulse of 250ms. The intensity will be varying according the painful threshold of each patient. After, the ischemic compression will be applied. For this we will use an algometer to get maximum of homogeneity on therapy. The pressure intensity will be placed by the average between the values gotten during three previously measurements of threshold pain in each patient. The therapy will be applied in trigger point three times (60 seconds each) with 30 seconds of rest between the applications.
  Interventions: Procedure: Ischemic compression

INTERVENTIONS:
Drug: lidocaine — Women randomized for this treatment was submitted to 2mL of lidocaine 0,5% without vasoconstrictor, directly and perpendicularly on trigger point. Patients received lidocaine injections once a week for 4 weeks
  Other Names: Lidocaine injection
  Arms: lidocaine injection
Procedure: Ischemic compression — Women randomized for treatment with ischemic compression will be first subjected to transcutaneal electrostimulation(TENS) for 30 minutes on trigger point to inhibit the painful stimulation. For this will be used 100 Hertz of frequency and pulse of 250ms. The intensity will be varying according the painful threshold of each patient. After, the ischemic compression will be applied. For this we will use an algometer to get maximum of homogeneity on therapy. The pressure intensity will be placed by the average between the values gotten during three previously measurements of threshold pain in each patient. The therapy will be applied in trigger point three times (60 seconds each) with 30 seconds of rest between the applications.
  Arms: Ischemic compression

SUMMARY:
Our hypothesis is that with comparison of effectiveness of two most common techniques of treatment for myofascial pain syndrome (injection of local anesthesia and ischemic compression) we could choice the most adequate to treat this disease. This way we could decrease the expenses with medicines, examinations, consultations and the time that women remains without a diagnosis and treatment.

DETAILED DESCRIPTION:
After evaluation and diagnostic confirmation, the patients will be randomized and submitted to the treatment with lidocaine injection or ischemic compression. Each treatment will be placed once a week, for four weeks. Women randomized for treatment with Ischemic compression, will be first subjected to transcutaneal electrostimulation(TENS), in order to receive analgesia on trigger point. The analgesia will be used to inhibit the painful stimulation. The device used for this will be the Dualpex 961, with 100 Hertz of frequency and pulse of 250ms. The intensity will be vary according the painful threshold of each patient. The electrostimulation will be made for 30 minutes. The electrodes will be applied around the trigger point. After analgesia, the ischemic compression will be applied. This therapy consists in a continuous pressure on trigger point. For this we will use one algometer to get maximum of homogeneity on therapy. The pressure intensity will be placed by the average between the values gotten during three previously measurements of threshold pain in each patient. This therapy will be applied three times with duration of 60 seconds each with a 30 seconds of rest between the applications. Injection of anesthesia: this therapy will be applied directly in trigger points with two mL of lidocaine 0.5% with needle of 22 gauges directly and perpendicularly in trigger point. The Evaluations for each treatment will be carried immediately before the randomization; In one month: immediately after the four weeks of treatment; - Three months: three months after the treatment; - Six months: six months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women with chronic diagnosis of pelvic pain;
2. Women in menacme;
3. Presence of the diagnostic criteria for abdominal myofascial syndrome;
4. Agreement with the Term of Free and Clarified Assent.

Exclusion Criteria:

1. Endometriosis, interstitial cystitis, syndrome of the irritable intestine or another illness that it justifies or it contributes for chronic pelvic pain;
2. Endometrioma or hernia evidenced to the ultrasound of the abdominal wall.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2009-10 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omero Poli, doctor, Study Director — University of Sao Paulo
Locations (1):
- Center of Chronic Pelvic Pain and Gynecologic Endoscopy of Ribeirao Preto Medical School, University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Montenegro ML, Braz CA, Rosa-e-Silva JC, Candido-dos-Reis FJ, Nogueira AA, Poli-Neto OB. Anaesthetic injection versus ischemic compression for the pain relief of abdominal wall trigger points in women with chronic pelvic pain. BMC Anesthesiol. 2015 Dec 1;15:175. doi: 10.1186/s12871-015-0155-0. PMID 26628263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited at Center of Chronic Pelvic Pain at Hospital das Clinicas of Ribeirão Preto Medical School, during 2010. The study was early stopped because the comparator (lidocaine injection) appears significantly more effective.
Groups:
- TENS Plus Ischemic Compression: Group received TENS plus ischemic compression
- Anesthesia Injection: Group received lidocaine injection
Period: Overall Study
Arm/Group | TENS Plus Ischemic Compression | Anesthesia Injection
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ischemic Compression: Group received TENS plus Ischemic compression
- Anesthesia Injection: group received lidocaine injections once a week for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Ischemic Compression | Anesthesia Injection | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
  <=18 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (3.2) | 38.5 (2.8) | 37.6 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Intensity of Pain
Description: The pain will measured by using the visual analogue scale, that is represented by a straight line of 100mm starting at "absence of pain" and ending at point "worst pain experienced or imagined".
Time Frame: immediately, 1, 3 months after treatment
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Ischemic Compression: Group received ischemic compression
Arm/Group | Ischemic Compression | Anesthesia Injection
Number analyzed (Participants) | 14 | 14
millimeters
  immediately after treatment | 52.7 (22.2) | 33.7 (29.2)
  1 month after treatment | 53.0 (17.4) | 27.1 (33.4)
  3 months after treatment | 50.8 (24.4) | 20.8 (26.0)

2. Primary Outcome: Clinical Response Rate
Description: We analyzed the clinical response rate considering significative reduction of 50% of visual analogue scale or significative subjective improvement.
Time Frame: immediately, 1, 3 months after treatment
Measure: Number; unit: percentage of participants
Arm/Group | TENS Plus Ischemic Compression | Anesthesia Injection
Number analyzed (Participants) | 14 | 14
percentage of participants
  immediately after treatment | 17.5 | 45.3
  1 month after treatment | 8.8 | 60.2
  3 months after treatment | 7.0 | 69.9

ADVERSE EVENTS:
Description: Periodic medical visits and phone calls.
Arm/Group | Ischemic Compression | Anesthesia Injection
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ischemic Compression (N=15) | Anesthesia Injection (N=15)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) — 3.4 and 5.1 centimeter of extension that resolved spontaneously within 4 and 6 weeks after, respectively

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No